CLINICAL TRIAL: NCT01199276
Title: An International, Multi-center, Randomized, Controlled Trial Evaluating The Effect of Xenon on Post-operative Delirium in Elderly Patients Undergoing Hip Fracture Surgery
Brief Title: Hip Fracture Surgery in Elderly Patients
Acronym: HIPELD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Air Liquide Santé International (Industry)
Collaborators: OptumInsight (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ALMED-08-C2-020
Record Dates: First submitted 2010-09-09; First posted 2010-09-10 (Estimated); Last update posted 2015-07-27 (Estimated); Status verified 2015-07

CONDITIONS: Delirium
Keywords: Delirium; Hip Fracture; Elderly
MeSH Terms: conditions — Delirium; Hip Fractures | interventions — Xenon; Sevoflurane

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Xenon (Experimental): 60%(1MAC)in oxygen (FiO2 = 0.35-0.45)
  Interventions: Drug: Xenon
- Sevoflurane (Active Comparator): 1.1-1.4% (1 MAC) in oxygen (FiO2 = 0.35-0.45) and medical air
  Interventions: Drug: Sevoflurane

INTERVENTIONS:
Drug: Xenon — Group A: xenon 60% (55%-65%)(1 MAC) in oxygen (FiO2 = 0.35-0.45)
  Other Names: LENOXe
  Arms: Xenon
Drug: Sevoflurane — Group B: sevoflurane 1.1-1.4%(1 MAC) in oxygen (FiO2 = 0.35-0.45) and Medical air
  Arms: Sevoflurane

SUMMARY:
The objective of this study is to evaluate the incidence of Post-Operative Delirium (POD), diagnosed with the Confusion Assessment Method (CAM), in elderly patients undergoing hip fracture surgery under general anaesthesia with xenon or sevoflurane, for a period of four days post-surgery.

ELIGIBILITY:
Inclusion Criteria:

* Elderly patient (≥ 75 years)
* Patient with planned hip fracture surgery within 48 hours after the hip fracture
* Patient willing and able to complete the requirements of this study including the signature of the written informed consent

Exclusion Criteria:

* Patient suffering from multiple fractures, pelvic fractures proximal, pathological fractures, femur fractures (i.e., fractures of the middle or distal femur)
* Disabling neuropsychiatric disorders (severe dementia, Alzheimer's disease, schizophrenia, depression)
* Brain trauma within 12 months prior to selection, history of stroke with residuals
* Patient suffering from delirium (CAM diagnosis) at selection
* Patient who cannot complete the pre-operative mental tests (CAM and/or MMSE) of this clinical trial
* Patient with Mini-Mental State Examination (MMSE) score < 24 at selection
* Patient known to susceptible to malignant hyperthermia
* Patient with elevated intra-cranial pressure
* Patient with a risk of high oxygen demand
* Patient with recent or ongoing myocardial infarction / damage
* Patient with severe cardiac failure, or patient with severe impaired left ventricular systolic function
* Patient with known severe lung and/or airway disease, or severe chronic respiratory insufficiency, or a sustained homecare oxygen therapy
* Contra-indication (serious illness or medical conditions) for general anaesthesia
* Known allergy or hypersensitivity to any drugs administered during this clinical trial
* Previous participation in this clinical trial
* Participation in another clinical trial within 4 weeks prior to selection
* History of alcohol or drug abuse or psychiatric disorders which would impair the understanding of the necessary information or render medically or legally unable to give written informed consent

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 256 (Actual)
Dates: Start 2010-09; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Post Operative Delirium diagnosed with the Confusion Assessment Method within four days post-surgery | Four days

SECONDARY OUTCOMES:
Post Operative Delirium diagnosed with the Confusion Assessment Method from day 5 post surgery to discharge from hospital | About 7 days
Sequential Organ Failure Assessment from day 1 to day 4 post-surgery | four days
Recovery Parameters | fifteen minutes
economic parameters | up to thirty days
Safety Parameters | Up to thirty days
  Serious Adverse Events, Adverse Events, laboratory parameters

CONTACTS AND LOCATIONS:
Overall Officials: Mark COBURN, MD, Study Chair — University Hospital Aachen - Germany; Robert SANDERS, MD, Study Chair — Imperial College London - UK; Rolf ROSSAINT, MD, Study Chair — University Hospital Aachen - Germany
Locations (13):
- UZ Leuven, Leuven, Belgium
- France (6):
  - Centre Hospitalier Universitaire de Grenoble, La Tronche
  - Centre Hospitalier Régional Universitaire de Montpellier, Montpellier
  - Groupe Hospitalier La Pitié-Salpêtriere, Paris
  - Groupe Hospitalier COCHIN, Paris
  - CHU Pontchaillou - Université de Rennes 1, Rennes
  - Centre Hospitalier Universitaire de Toulouse, Toulouse
- Germany (3):
  - University Hospital Aachen, Aachen
  - . Klinik für Anästhesiologie - Universitätsklinikum Düsseldorf, Düsseldorf
  - Klinikum Mutterhaus Der Borromaerinnen, Trier
- IRCCS Rizzoli Orthopaedic Institute, Bologna, Italy
- Hospital Clinico Universitario de Valencia, Valencia, Spain
- Imperial College NHS Trust, London, United Kingdom

REFERENCES:
- [Derived] Coburn M, Sanders RD, Maze M, Nguyen-Pascal ML, Rex S, Garrigues B, Carbonell JA, Garcia-Perez ML, Stevanovic A, Kienbaum P, Neukirchen M, Schaefer MS, Borghi B, van Oven H, Tognu A, Al Tmimi L, Eyrolle L, Langeron O, Capdevila X, Arnold GM, Schaller M, Rossaint R; HIPELD Study Investigators. The hip fracture surgery in elderly patients (HIPELD) study to evaluate xenon anaesthesia for the prevention of postoperative delirium: a multicentre, randomized clinical trial. Br J Anaesth. 2018 Jan;120(1):127-137. doi: 10.1016/j.bja.2017.11.015. Epub 2017 Nov 21. PMID 29397119
- [Derived] Coburn M, Sanders RD, Maze M, Rossaint R; HIPELD Investigators. The Hip Fracture Surgery in Elderly Patients (HIPELD) study: protocol for a randomized, multicenter controlled trial evaluating the effect of xenon on postoperative delirium in older patients undergoing hip fracture surgery. Trials. 2012 Sep 27;13:180. doi: 10.1186/1745-6215-13-180. PMID 23016882